CLINICAL TRIAL: NCT06300294
Title: Effect of Acupressure on Anxiety, Pain and Vital Signs in Individuals Diagnosed With Acute Coronary Syndrome: A Randomized Controlled Study
Brief Title: Acute Coronary Syndrome and Acupressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, ASSOCIATE PROFESSOR DOCTOR, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-AYN-3
Record Dates: First submitted 2024-02-14; First posted 2024-03-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome; Nursing
Keywords: acupressure, anxiety, vital signs, acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: experimental and control
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Since block randomization will be used in the study, the research director and the individuals who meet the study inclusion criteria will not know which group they will be in during the preliminary evaluation process of the study. However, the person analyzing the data will not know which group the data belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): acupressure application and Routine care and treatment (filling out the initial hospitalization documents, measuring vital signs, taking an ECG, preparing for the CAG procedure, administering the ordered medications).
  Interventions: Other: acupressure
- control (No Intervention): Routine care and treatment (filling out the initial hospitalization documents, measuring vital signs, taking an ECG, preparing for the CAG procedure, administering the ordered medications).

INTERVENTIONS:
Other: acupressure — After the CAG procedure, acupressure will be applied to individuals whose vital signs are within the normal range.
  Arms: acupressure

SUMMARY:
This study aims to examine the effect of acupressure on physiological parameters and anxiety levels in individuals diagnosed with Acute Coronary Syndrome (ACS).

H1-1: Acupressure applied to individuals diagnosed with ACS has an effect on the level of anxiety.

H1-2: Acupressure applied to individuals diagnosed with ACS has an effect on blood pressure.

H1-3: Acupressure applied to individuals diagnosed with ACS has an effect on heart rate.

H1-4: Acupressure applied to individuals diagnosed with ACS has an effect on respiratory rate.

H1-5: Acupressure applied to individuals diagnosed with ACS has an effect on the pain level.

H1-6: Acupressure applied to individuals diagnosed with ACS has an effect on cortisol levels.

DETAILED DESCRIPTION:
Acute Coronary Syndrome (ACS) affects millions of people every year; It refers to three types of coronary artery disease: unstable angina pectoris, non-ST-elevation myocardial infarction (NSTE MI) and ST-elevation myocardial infarction (STEMI). It is known that 19 million people in the world and 161 thousand people in our country lost their lives due to Cardiovascular Disease (CVD). Approximately 3 million people worldwide die due to STEMI.Individuals experiencing ACS generally; It is observed that he/she experiences burning, stinging and compressive chest pain, tachycardia, sweating, fatigue, dizziness, dyspnea, nausea, anxiety and depression.Management of the disease is combined with pharmacological applications; It is tried to be provided with non-pharmacological applications such as education, acupuncture and acupressure. When the literature is examined, acupressure application; in the physiological parameters of individuals with myocardial infarction; It brings blood pressure, heart rate and respiratory rate to normal limits, and increases oxygen saturation and sleep quality; It appears to reduce anxiety and pain.For all these reasons, this study aims to examine the effect of acupressure on physiological parameters (blood pressure, heart rate, respiratory rate, pain and cortisol) and anxiety levels in individuals diagnosed with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,

  * Those aged 18 and over
  * Able to speak Turkish
  * Diagnosed with ACS for the first time
  * Cardiopulmonary resuscitation not applied
  * No orientation problems (those who score 15 on the Glasgow Coma Scale)
  * Not diagnosed with psychiatric disease
  * No amputation, fistula, lymphedema, neuropathy or hemiplegia in any of the Upper Extremities
  * Those who underwent femoral intervention for CAG procedure
  * Those who have not used any integrative practices based on pressure and stimulation such as acupressure, acupuncture and reflexology in the last month.
  * Vital signs (28) are within normal range:

Blood pressure: 90/60-120/80 mmHg Heart rate: 60-100 min Respiratory rate: 12-18 min

Exclusion Criteria:

* Those with arrhythmia (AF, VT etc.)
* Patients who have previously undergone Coronary Angiography
* Diagnosed with myocarditis, pericarditis
* Those who do not take any speed-breaking drugs (beloc, arlec, etc.).
* Patients who underwent radial intervention for CAG procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
means of blood pressure | up to 30 minutes
  In this study, blood pressure was measured using monitors in the intensive care unit.
means of hear rate | up to 30 minutes
  Heart rate is the pressure exerted on the vessel wall by the blood thrown by the left ventricle from the skin surface to the aorta during systole. In the research, heart rate is measured using a monitor.
means of respiratory rate | up to 30 minutes
  Respiratory rate is the patient's breaths per minute. In this study, respiratory rate was taken from the monitor.
means of cortisol. | up to 60 minutes
  The cortisol value in the blood will be measured.

SECONDARY OUTCOMES:
means of subjective anxiety scores. | up to 30 minutes
  numerical anxiety scale. The total score between 0-10 obtained.
means of subjective pain scores. | up to 30 minutes
  visual analog scale. It consists of a straight line with endpoints that define end limits such as "no pain" and "pain as bad as possible". The patient is asked to mark the level of pain on the line between the two endpoints.
electrocardiography evaluation | up to 30 minutes
  Electrocardiography is the process of recording the electrical activity occurring in the heart to examine the functioning of the heart muscle and neural conduction system.

CONTACTS AND LOCATIONS:
Overall Officials: aynur açıkgöz, PhD student, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Manisa City Hospital, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No